CLINICAL TRIAL: NCT02757222
Title: Intensifying Radiation Treatment in Advanced/ Poor Prognosis Laryngeal, Hypopharyngeal (LH) and Oropharyngeal Cancers (OPC) Using PET -CT Based Dose Escalation Strategies ( INTELHOPE)
Brief Title: Dose Escalation Versus Standard in Laryngopharyngeal Cancers
Acronym: INTELHOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/TMC/38/14
Record Dates: First submitted 2016-03-22; First posted 2016-05-02 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Malignant Neoplasm of Oropharynx Stage III; Malignant Neoplasm of Larynx Stage III; Malignant Neoplasm of Hypopharynx Stage III; Malignant Neoplasm of Oropharynx Stage IVa; Malignant Neoplasm of Oropharynx Stage IVb; Malignant Neoplasm of Larynx Stage IV; Malignant Neoplasm of Hypopharynx Stage IVa; Malignant Neoplasm of Hypopharynx Stage IVb
MeSH Terms: conditions — Oropharyngeal Neoplasms; Laryngeal Neoplasms; Hypopharyngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: It is a radiation dose escalation study.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard dose (Active Comparator): Patients receive a radiation dose of 66Gy in 30 fractions to the planning target volume 1 (PTV1) and 54 Gy in 30 fractions to the PTV2 concurrent with platinum chemotherapy weekly
  Interventions: Radiation: Standard Dose
- Escalated dose (Experimental): Patients receive a radiation dose of 73.5 Gy in 30 fractions to the boost target volume (BTV), 63Gy in 30 fractions to PTV1 and 54 Gy in 30 fractions to PTV2 concurrent with platinum chemotherapy weekly
  Interventions: Radiation: Escalated Dose

INTERVENTIONS:
Radiation: Escalated Dose — Boost Target Volume (BTV): The PET CT GTV (thresholding at 40% of SUV max) with a 3mm margin will form the BTV.
  CTV1: A 3mm area around the BTV avid primary or 2mm area around the node will form the CTV1.
  CTV 2: This (CTV 2) includes the area around the primary or nodal levels at risk of harbouring microscopic primary or microscopic nodal metastatic disease and not already included in CTV1.
  Planning Target Volume: PTV - A margin of 5mm will be added to each of the CTV to obtain the PTV.
  BTV receives 73.5Gy in 30 fractions. PTV 1 receives 63Gy in 30 fractions. PTV 2 receives 54 Gy in 30 fractions.
  All patients receive concurrent platinum chemotherapy.
  Arms: Escalated dose
Radiation: Standard Dose — CTV 1 includes 6mm isotropic margin around the entire PET-CT avid (thresholding at 40% of SUV max) larynx/ hypopharynx /oropharynx and 5mm isotropic margin around nodes.
  CTV 2: This (CTV 2) includes the area around the primary or nodal levels at risk of harbouring microscopic primary or microscopic nodal involvement, or at risk nodal areas, and not already included in CTV1.
  Planning Target Volume: PTV - A margin of 5mm will be added to each of the CTV to obtain the PTV.
  PTV 1 receives 66Gy in 30 fractions. PTV 2 receives 54 Gy in 30 fractions.
  All patients receive concurrent platinum chemotherapy.
  Arms: Standard dose

SUMMARY:
The primary objective of the study is to establish the safety of using a moderate escalation of radiotherapy dose in advanced/poor prognosis OPC and LH cancers receiving curative radiotherapy.

The study will also explore the efficacy (improvement in complete response rates at 2 years) of dose escalation in intermediate and high risk OPC and LH cancers patients.

DETAILED DESCRIPTION:
Patients with locally advanced Laryngeal, Hypopharyngeal (LH) or oropharyngeal (OPC) head and neck squamous cell carcinomas have 5 year survival ranging between 25-45%. 60% of all LH cancers occur in the developing world and its incidence in India ranges from 1.8-8.8 per 1,00,000 population .

Local control outcomes of OPC patients with stage III and IV OPC has been modest with reported loco-regional control rates of 50-60% at 5 years. For patients with locally advanced LH a 60-70% 2 year survival is seen and loco-regional control rates of 70% have been reported . Majority of locally advanced OPC and LH cancers are treated with a combination of chemotherapy and radiotherapy (CRT) with organ and function preserving approach.

Identifying the area of tumour involvement in the OPC and LH could be challenging on CECT scans, requiring metabolic imaging with PET-CT for more precise definition of radiation target.

Improvements in radiation treatment delivery techniques have enabled clinicians to explore the possibility of improving tumour control probability (TCP) and reduce normal tissue complication probability . This allows us to explore the role of escalating dose in the above group of patients to assess the safety and efficacy of the regime.

Tumours treated in the standard dose arm will receive radiotherapy @ 220 cGy per fraction for 30 fractions whilst those in the escalated dose arm will receive @ 245 cGy per fraction for 30 fractions using IMRT techniques. Patients in both arms will receive weekly platinum based chemotherapy concurrent with radiotherapy.

ELIGIBILITY:
LH Inclusion Criteria ALL of the following inclusion criteria must be met

* Histologically confirmed squamous cell cancer of the larynx or hypopharynx
* Radiotherapy with concomitant chemotherapy as primary therapy
* Induction chemotherapy is permitted
* TNM Stage T3-4, N0-3, M0 or T1/2 with N2-3 disease (Stage III or IV a/b) disease
* WHO performance status of 0 or 1
* Creatinine clearance of more than 50ml/min
* All patients must be suitable to attend regular follow up

OPC inclusion criteria ALL of the following inclusion criteria must be met

* Histologically confirmed squamous cell cancer of the oropharynx
* Radiotherapy with concomitant chemotherapy as primary therapy
* Induction chemotherapy is permitted
* WHO performance status of 0 or 1
* Creatinine clearance of more than 50ml/min
* All patients must be suitable to attend regular follow up
* And any of the stage of disease as seen below HPV (p16) negative: TNM Stage T2-T4, any N stage, M0 disease HPV (p16) Positive: more than 10 pack year history and N2b or N3 disease

LH Exclusion Criteria The patient is ineligible if ANYONE of the following exclusion criteria is met

* Previous radiotherapy to the head and neck region
* Previous malignancy except non-melanoma skin cancer and early stage cancer in remission for at least 5 years following treatment
* Previous or concurrent illness, which in the investigator's opinion would interfere with either completion of therapy or follow-up
* Pre-existing previous speech or swallowing problems unrelated to the diagnosis of cancer
* Patients with locally advanced LH tumours where organ preservation is unrealistic
* Patients with metastatic carcinoma

OPC Exclusion Criteria The patient is ineligible if ANYONE of the following exclusion criteria is met

* Previous radiotherapy to the head and neck region
* Previous malignancy except non-melanoma skin cancer and early stage cancer in remission for at least 5 years following treatment
* Previous or concurrent illness, which in the investigator's opinion would interfere with either completion of therapy or follow-up
* Pre-existing previous speech or swallowing problems unrelated to the diagnosis of cancer
* Patients with locally advanced LH or OPC tumours where organ preservation is unrealistic
* Patients with metastatic carcinoma
* Low risk OPC: HPV p16 positive T1-2 with N0-N2a disease or less than 10 pack year history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with Grade 3 through grade 5 adverse events that are related to dose escalation, graded according to NCI CTCAE version 4.0 | 2 years
  In addition: Interim assessment for early stoppage is if 35% or more patients in the intervention arm has Grade 4 mucositis or dysphagia

SECONDARY OUTCOMES:
Efficacy (improvement in complete response rates at 2 years) of dose escalation in intermediate and high risk Oropharyngeal cancer (OPC) patients and in node positive, locally advanced Laryngeal and Hypopharyngeal cancer patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sanjoy Chatterjee, FRCP, FRCR, Principal Investigator — Tata Medical Center: Kolkata
Locations (1):
- Tata Medical Centre, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: Undecided
Once appropriate authorities approach and once clearance of local authorities is received, data could be shared

REFERENCES:
- [Background] Kapil U, Singh P, Bahadur S, Dwivedi SN, Singh R, Shukla N. Assessment of risk factors in laryngeal cancer in India: a case-control study. Asian Pac J Cancer Prev. 2005 Apr-Jun;6(2):202-7. PMID 16101334
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Background] Chatterjee S, Willis N, Locks SM, Mott JH, Kelly CG. Dosimetric and radiobiological comparison of helical tomotherapy, forward-planned intensity-modulated radiotherapy and two-phase conformal plans for radical radiotherapy treatment of head and neck squamous cell carcinomas. Br J Radiol. 2011 Dec;84(1008):1083-90. doi: 10.1259/bjr/53812025. PMID 22101580
- [Result] Guerrero Urbano T, Clark CH, Hansen VN, Adams EJ, A'Hern R, Miles EA, McNair H, Bidmead M, Warrington AP, Dearnaley DP, Harrington KJ, Nutting CM. A phase I study of dose-escalated chemoradiation with accelerated intensity modulated radiotherapy in locally advanced head and neck cancer. Radiother Oncol. 2007 Oct;85(1):36-41. doi: 10.1016/j.radonc.2007.07.011. Epub 2007 Aug 20. PMID 17709149
- [Result] Overgaard J, Hansen HS, Specht L, Overgaard M, Grau C, Andersen E, Bentzen J, Bastholt L, Hansen O, Johansen J, Andersen L, Evensen JF. Five compared with six fractions per week of conventional radiotherapy of squamous-cell carcinoma of head and neck: DAHANCA 6 and 7 randomised controlled trial. Lancet. 2003 Sep 20;362(9388):933-40. doi: 10.1016/s0140-6736(03)14361-9. PMID 14511925
- [Result] Fu KK, Pajak TF, Trotti A, Jones CU, Spencer SA, Phillips TL, Garden AS, Ridge JA, Cooper JS, Ang KK. A Radiation Therapy Oncology Group (RTOG) phase III randomized study to compare hyperfractionation and two variants of accelerated fractionation to standard fractionation radiotherapy for head and neck squamous cell carcinomas: first report of RTOG 9003. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):7-16. doi: 10.1016/s0360-3016(00)00663-5. PMID 10924966
- [Result] Leclerc M, Maingon P, Hamoir M, Dalban C, Calais G, Nuyts S, Serre A, Gregoire V. A dose escalation study with intensity modulated radiation therapy (IMRT) in T2N0, T2N1, T3N0 squamous cell carcinomas (SCC) of the oropharynx, larynx and hypopharynx using a simultaneous integrated boost (SIB) approach. Radiother Oncol. 2013 Mar;106(3):333-40. doi: 10.1016/j.radonc.2013.03.002. Epub 2013 Mar 27. PMID 23541643
- [Result] Paleri V, Carding P, Chatterjee S, Kelly C, Wilson JA, Welch A, Drinnan M. Voice outcomes after concurrent chemoradiotherapy for advanced nonlaryngeal head and neck cancer: a prospective study. Head Neck. 2012 Dec;34(12):1747-52. doi: 10.1002/hed.22003. Epub 2012 Feb 9. PMID 22319013